CLINICAL TRIAL: NCT05117775
Title: Towards A Better Paradigm for Head and Neck Cancer Treatment Applying Artificial Intelligence: an International Cohort Study of Electronic Health Records. HNC-TACTIC.
Brief Title: Towards A Better Paradigm for Head and Neck Cancer Treatment Applying Artificial Intelligence. HNC-TACTIC.
Acronym: HNC-TACTIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Savana Research (Network)
Collaborators: Head and Neck Cancer International Group (HNCIG) (Unknown)
Responsible Party: Sponsor
Other Study IDs: HNC-TACTIC
Record Dates: First submitted 2021-10-08; First posted 2021-11-11 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Head and Neck Cancer
Keywords: HNSCC; Predictive factors; Overall survival; Immunotherapy; Electronic health records; Natural language processing; Artificial intelligence
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with all stages of HNSCC (Full analysis set): To describe median OS by primary tumor location (oral cavity, oropharynx, larynx, and hypopharynx) in HNSCC patients after stratification for prognostic factors, including tumor stage and treatment.
  Interventions: Other: No intervention - Just description and predictive models
- Patients with early and locally advanced stages: To describe clinical characteristics and treatments and to compare OS in locally advanced HNSCC patients
  Interventions: Other: No intervention - Just description and predictive models
- Patients with recurrent or metastatic disease: To describe the epidemiologic and clinical characteristics, and treatment and the impact of introducing immunotherapy in recurrent or metastatic HNSCC
  Interventions: Other: No intervention - Just description and predictive models

INTERVENTIONS:
Other: No intervention - Just description and predictive models — All the groups will be descriptive, there is not intervention, as it is an Observational study applying artificial Intelligence (RWE).

SUMMARY:
This will be an international, multicenter, retrospective, observational, and data-driven study using secondary data captured in EHRs. The extraction of the data captured in the EHRs will be performed with SAVANA's EHRead®, an innovative data-driven system based on Natural Language Processing (NLP) and machine learning. For all patients, the Index Date is defined as the timepoint within the study period when they fulfill ALL inclusion criteria and no exclusion criteria. Follow-up comprises the period between Index Date and the last EHR available within the study period. Additional variable-specific time windows may be considered to optimize data collection.

DETAILED DESCRIPTION:
The present study aims to describe the clinical characteristics of patients with HNSCC in a real-world setting by analyzing readily available information in the Electronic Health Records (EHRs). This study will gain a deep insight of the clinical characteristics and real-world outcomes of patients with all stages (early, locally advanced, and metastatic) of HNSCC. It will focus on developing two predictive models to apply in the clinical setting, one for electing patients with high-risk of recurrence after radical treatment, and the second one for selecting recurrent or metastatic patients who could benefit from immunotherapy.

To achieve the proposed study objectives we will use SAVANA´s EHRead® (11-15), a technology that applies Natural Language Processing (NLP) (16) and machine learning to extract, organize, and analyze the unstructured clinical information jotted down by health professionals in patients' EHRs.

Primary objectives

* To develop a predictive model based on dynamic risk stratification (DRS) for the risk of recurrence or disease progression following a primary curative treatment in HNSCC patients with early and locally advanced disease.
* To develop a predictive model based on dynamic risk stratification (DRS) aimed at identifying patients' features that predict long-term survival after immunotherapy in recurrent and metastatic HNSCC patients. Secondary objectives
* To describe median OS by primary tumor location (oral cavity, oropharynx, larynx, and hypopharynx) in HNSCC patients after stratification for prognostic factors, including tumor stage and treatment.
* To describe the demographics, clinical characteristics, and treatment of patients with HNSCC in early and locally advanced stages of the disease.
* To describe the patterns of follow-up in patients with HNSCC in early and locally advanced stages of the disease.
* Departments in charge
* Number of visits
* Imaging and anatomopathological tests
* Recurrence detected by physical examination.
* To evaluate the impact of treatments on patients with locally advanced stages of the disease.
* Patients' early and late toxicity to the treatment, comparing between radiotherapy (+/-cisplatin or cetuximab) vs surgery and post-operative r< radiotherapy (+/- cisplatin).
* Healthcare resource utilization (HCRU), including medical visits, diagnostics, and hospitalizations.
* To compare OS in locally advanced HNSCC patients (including both HPV+ and HPV- oropharyngeal patients) treated with cisplatin-radiotherapy vs cetuximab-radiotherapy and treated with surgery vs. conservative treatment.
* To compare the demographic and clinical characteristics of exceptional responders and poor responders (based on recurrence and long-term survival). This analysis will be performed independently for HPV+ and HPV- oropharyngeal patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old.
* Patients diagnosed with HNSCC
* For selected exploratory analyses, patients diagnosed with nasopharynx, paranasal sinus, and salivary gland tumors.

Exclusion Criteria:

* Patients with follow-up of less than 6 months, except if deceased (any cause) in the 6 months after HNSCC diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Full Analysis Set (FAS) will comprise all adult patients with all stages of HNSCC. For completion of secondary objectives, two different subgroups based on stage of the disease will be considered. Treatment approaches will be analyzed in different cohorts of patients within each subgroup.
  * Partial Analysis Set (PAS) 1: Patients with early stages of the disease
  * PAS 2.1: Patients with locally advanced stages of the disease diagnosed with HPV-negative HNSC.
  * PAS 2.2: Patients with locally advanced stages of the disease diagnosed with HPV-positive oropharyngeal squamous cell carcinoma.
  * PAS 3: Patients with recurrent/metastatic disease.
  * PAS 4 (for exploratory analysis): Patients diagnosed with nasopharynx, paranasal sinus, and salivary gland tumors.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive model based on dynamic risk stratification (DRS) for the risk of recurrence or disease progression | From 1st Jan 2021
  To develop a predictive model based on dynamic risk stratification (DRS) for the risk of recurrence or disease progression following a primary curative treatment in HNSCC patients with early and locally advanced disease.
Predictive model based on dynamic risk stratification (DRS) aimed at identifying patients' features | From 1st Jan 2021
  To develop a predictive model based on dynamic risk stratification (DRS) aimed at identifying patients' features that predict long-term survival after immunotherapy in recurrent and metastatic HNSCC patients

SECONDARY OUTCOMES:
In all patients with all stages of HNSCC (full analysis set, FAS): | From 1st Jan 2021
  To describe median OS by primary tumor location (oral cavity, oropharynx, larynx, and hypopharynx) in HNSCC patients after stratification for prognostic factors, including tumor stage and treatment.
In patients with early and locally advanced stages of the disease (including all patients treated with curative intent): | From 1st Jan 2021
  * To describe the demographics, clinical characteristics, and treatments
  * To describe the patterns of follow-up
  * Departments in charge
  * Number of visits
  * Imaging and anatomopathological tests
  * Recurrence detected by physical examination
  * To evaluate the impact of treatments on patients with locally advanced stages of the disease.
  * Patients' early and late toxicity to the treatment, comparing between radiotherapy (cisplatin or cetuximab) vs surgery and post-operative radiotherapy (cisplatin)
  * Healthcare resource utilization (HCRU), including medical visits, diagnostics, and hospitalizations.
  * To compare OS in locally advanced HNSCC patients (including both HPV+ and HPV- oropharyngeal patients) treated with cisplati
In patients with recurrent or metastatic disease: | From 1st Jan 2021
  * To describe the epidemiologic and clinical characteristics, and treatments
  * To describe epidemiologic, clinical, and tumor characteristics of long-term survivors treated with immunotherapy and non-immunotherapy approaches.
  * To describe the impact of introducing immunotherapy in recurrent or metastatic
  HNSCC:
  * Treatment outcome: OS
  * HCRU, including medical visits, diagnostics, and hospitalizations.

OTHER OUTCOMES:
Exploratory objective | From 1st Jan 2021
  To describe the demographics, clinical characteristics, and treatment of patients with nasopharynx, paranasal sinus, and salivary gland tumors.

CONTACTS AND LOCATIONS:
Overall Officials: John Almeida, Study Chair — University Health Network and Mount Sinai Hospital; Sujith Baliaga, Study Chair — Ohio State University; David Casadevall, Study Chair — Medsavana S.L; Melvin Chua, Study Chair — National Cancer Centre, Singapore; Andreas Dietz, Study Chair — University Hospital of Leipzig; Robert Ferris, Study Chair — UPMC Hillman Cancer Center; Raul Giglio, Study Chair — Hopital Ángel H. Roffo de Buenos Aires; Chris Holsinger, Study Chair — Stanford University; Kate Hutcheson, Study Chair — M.D. Anderson Cancer Center; Husham Menhanna, Study Chair — Institute of Head and Neck Studies and Education (InHANSE); Pablo Parente, Study Chair — Hospital HM Rosaleda; Sandro Porceddu, Study Chair — Queensland Institute of Medical Research (QIMR); Miren Taberna, Principal Investigator — Medsavana S.L; Christian Simon, Study Chair — CHUV Lausanne
Locations (1):
- Savan Research S.L, Madrid, Spain